CLINICAL TRIAL: NCT05522985
Title: A Single Center, Prospective, Randomized Controlled, Phase II Clinical Study of Anti-PD-1 Antibody js001 (Treprizumab) Combined With TP Neoadjuvant Chemotherapy in the Treatment of Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant Chemotherapytreatment of Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCIHMF&ENT-002
Record Dates: First submitted 2022-08-09; First posted 2022-08-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Chemotherapy
Keywords: Head and neck squamous cell carcinoma; Neoadjuvant chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treprizumab combined with TP (Experimental): treprizumab injection: 240mg once, intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.
  paclitaxel for injection (albumin binding type) 260 mg / m2, intravenous drip, D1, every 3 weeks as a cycle, a total of 3 cycles; cisplatin: 75mg / m2, intravenous drip, D1, once every 3 weeks, a total of 3 cycles; Treprizumab was infused before and at least 60 minutes apart from chemotherapy; The intravenous infusion time of treprizumab shall be at least 60 minutes. Intravenous bolus or single rapid intravenous injection is not allowed.
  Interventions: Drug: Triprilimab combined with TP
- TP（paclitaxel +cisplatin） (Active Comparator): paclitaxel for injection (albumin binding type) 260 mg / m2, intravenous drip, D1, every 3 weeks as a cycle, a total of 3 cycles; cisplatin: 75mg / m2, intravenous drip, D1, once every 3 weeks, a total of 3 cycles;
  Interventions: Drug: Triprilimab combined with TP

INTERVENTIONS:
Drug: Triprilimab combined with TP — Both interventions all drugs intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.

SUMMARY:
The objective of research is to evaluate the efficacy and safety of treprizumab injection combined with AP regimen in the treatment of resectable locally advanced head and neck squamous cell carcinoma.122 patients were randomly divided into two groups: the test group (treprizumab injection combined with AP protocol) and the control group (TP protocol); The patients in both groups were treated with three cycles of induction therapy. After the induction therapy, the patients were evaluated and followed up with surgery.

DETAILED DESCRIPTION:
The case report form shall be filled by the investigator, and each selected case must complete the case report form. The completed case report form is used for data entry and management.

All original data were retained by the research department.Full analysis set: according to the principle of intention to analyze (ITT), all cases who received drug treatment and took drugs at least once were analyzed for efficacy. For the case data that cannot observe the whole treatment process, the last observation data shall be carried forward to the final results of the study (LOCF).

Per-protocol set: all cases that comply with the study protocol, have good compliance, have not taken prohibited drugs during the study period, and have completed the contents specified in the case report form. No imputation was performed for missing data. Fas and PPS were analyzed statistically for the efficacy of the drug.

Safety analysis set: all enrolled patients who have used the study drug at least once and have safety records after drug use belong to the safety analysis set. This data set was used for safety analysis.

All statistical analysis will be calculated by SPSS statistical analysis software. All statistical tests are conducted by two-sided test. If the p value is less than or equal to 0.05, the difference tested will be considered statistically significant. The confidence interval is 95%.

Baseline data were analyzed according to the full analysis set, and all efficacy indicators were analyzed according to the full analysis set and the compliance scheme set; The safety analysis set is adopted for the safety analysis.

Sample size calculated by PASS 11.0 software: According to the existing literature reports, the PCR rate of neoadjuvant therapy for locally advanced squamous cell carcinoma of the head and neck is about 16%. It is expected that the combined treatment with toripalimab can increase it to 40%. The sample size was calculated using the Test for Two Proportion sample size calculation module in the PASS software, with P1 set at 40% and P2 at 16%. Bilateral α=0.05, β=0.2. After calculation, the probability of a 24% difference between the detection groups was 80.743%. The sample size for both groups was 52 cases, with a total of 104 cases enrolled. The dropout rate was expected to be 15%, and the final sample size was 122 cases.

ELIGIBILITY:
Inclusion Criteria：

* The subject has head and neck squamous cell carcinoma confirmed by histopathology or cytology.
* Resectable, clinical stage III or IV and no distant metastasis (AJCC 8th)
* Initial treatment patients who have not received chemotherapy, radiotherapy, immunotherapy or biological therapy.
* There is at least one measurable lesion (RECIST 1.1 standard, see Annex 1).
* ECoG score: 0-1.
* Expected survival time ≥ 3 months.
* The functions of important organs meet the following requirements (no blood component, cell growth factor, white blood medicine, platelet medicine and anemia correction medicine are allowed to be used within 14 days before the first use of the study drug);WBC≥3.0x109 /L，ANC≥2.0x109/L,HB≥90g/L, Platelets ≥ 100x109 / L,Serum albumin ≥ 2.8g/dl,Total bilirubin ≤ 1.5xuln, ALT and AST ≤ 3.0xuln,Serum creatinine ≤ 1.5xuln or creatinine clearance rate > 60ml / min (Cockcroft Gault, see Appendix 4),Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5xuln (for anticoagulant therapy using stable doses such as low molecular weight heparin or warfarin and INR can be screened within the expected therapeutic range of anticoagulants)
* No contraindications of chemotherapy and immunotherapy.
* No history of immune related diseases.
* No uncontrollable pneumonia and pulmonary infection.
* Subjects of childbearing age must agree to take effective contraceptive measures during the trial; The serum or urine pregnancy test of women of childbearing age 72 hours before the start of chemotherapy must be negative.
* The subject has good compliance, can carry out treatment and follow-up, and voluntarily complies with the provisions of this study.
* The subjects voluntarily signed informed consent. Exclusion Criteria
* Patients with distant metastasis.
* There are uncontrolled serious medical diseases, such as complicated serious medical diseases, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
* Patients with a history of allergy or allergic constitution to any component of monoclonal antibody drugs in the past.
* Uncontrollable cardiac clinical symptoms or diseases, such as heart failure above NYHA grade II or left ventricular ejection fraction (LVEF) < 50% indicated by color Doppler echocardiography; Unstable angina pectoris; Myocardial infarction occurred within 1 year; Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention (including QTc interval ≥ 470 MS);
* Serious infection (CTC AE > grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia and infection complications requiring hospitalization; Baseline chest imaging revealed active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of study drug, or the need for oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics).
* Unexplained fever > 38.5 ° C occurred during the screening period and before the first administration (tumor fever can be included in the group according to the judgment of the investigator);
* Active autoimmune diseases and history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism and hypothyroidism, including but not limited to these diseases or syndromes); But does not include autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes using a stable dose of insulin; Patients with vitiligo or childhood asthma / allergy who have been cured and do not need any intervention after adulthood;
* Have a history of immune deficiency, including HIV test positive, or have other acquired and congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation.
* Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU / ml, or patients with active hepatitis C virus (HCV) should be excluded; Inactive hepatitis B surface antigen carriers, treated and stable hepatitis B patients (HBV DNA < 500iu / ml), and cured hepatitis C patients can be included in the group.
* Have a history of interstitial lung disease (excluding radiation pneumonia without hormone treatment) and non-infectious pneumonia.
* Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year before but without formal treatment.
* Patients who have received any of the following treatments;1)Received any investigational drug within 4 weeks before the first use of investigational drug; 2) Receive the last dose of anticancer treatment (including chemotherapy, radiotherapy, targeted therapy, etc.) within 4 weeks before the first use of the study drug;3)Subjects who need to be given corticosteroids (> 10 mg prednisone equivalent dose per day) or other immunosuppressants for systemic treatment within 2 weeks before the first use of the study drug, except for the use of corticosteroids for local inflammation and prevention of allergy, nausea and vomiting. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenocortical hormone replacement at doses > 10 mg / day prednisone efficacy dose were allowed ;4) Those who have been vaccinated with anti-tumor vaccine or have been vaccinated with live vaccine within 4 weeks before the first administration of the study drug; 5) Major surgery or severe trauma within 4 weeks before the first use of study drug; 6) Another clinical study was also included.
* There is dementia, mental state change or any mental illness that will hinder understanding or making informed consent or filling out questionnaires.
* subjects with ≥ grade 2 peripheral neuropathy according to CTCAE V5.0;
* History of allergy or hypersensitivity to any therapeutic ingredient.
* Primary malignant tumors other than head and neck squamous cell carcinoma in the past 5 years, except for fully treated basal cell or squamous epithelial cell skin cancer, local prostate cancer after radical operation, and ductal carcinoma in situ after radical operation.
* Those who need to be treated with other anti-tumor drugs.
* The investigator thinks that it is not suitable for enrollment.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2027-11-07 (Estimated)

PRIMARY OUTCOMES:
PCR | 9 weeks
  Pathological complete response rate

SECONDARY OUTCOMES:
MPR | 9 weeks
  major pathological remission

OTHER OUTCOMES:
ORR | 9 weeks
  objective response rate
OS | 2 years
  overall survival
PFS | 2 years
  progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China